CLINICAL TRIAL: NCT02766569
Title: International Registry for Secundum Atrial Septal Defects Closure by Using the Occlutech®Flex II Device in More Than 2000 Patients
Brief Title: International Registry for ASD Closure by Using the Occlutech®Flex II Device in More Than 2000 Patients
Acronym: IRFACODE-II
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. Nikolaus Haas, MD, PhD, FRACP, Prof. Dr. Nikolaus A. Haas, Ludwig-Maximilians - University of Munich
Other Study IDs: IRFACODE II
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Septal Defect
Keywords: IRFACODE II, ASD closure, ASD device, erosion, arrhythmia
MeSH Terms: conditions — Heart Septal Defects, Atrial; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ASD closure with the Occlutech Flex II ASD closure device — Monitoring of possible device related side effects with a minumum of 1 year follow-up.

SUMMARY:
The IRFACODE II study will evaluate the performance and safety of the Occlutech® Flex II device in patients with closure of secundum atrial septal defects (ASD II).

DETAILED DESCRIPTION:
Introduction: Interventional ASD closure is generally a safe procedure with only a small amount of severe side effects including mainly erosion of the atrial wall, embolizations and arrhythmias. The IRFACODE study has shown excellent results in Patients with various generations of the Occlutech devices. IRFACODE II study will evaluate the performance and safety of the Occlutech® Flex II device in patients with closure of secundum atrial septal defects (ASD II).

Methods: The IRFACODE II study is a retrospective, non-randomized open access study for centres with a minimum of about 50 patients to evaluate the safety and side effects of ASD closure with this device. A minimum of 2000 patients that have an ASD II closed with this device until 31. June 2016 will be enrolled, the follow-up will be until 31. June 2017. Primary outcome measures for safety are the amount of erosions over a minimum follow-up time of 12 months. Primary outcome measures for device performance will include the success of complete ASD closure. Secondary outcome measures for safety will include the technique of implantation, the success rate in anatomically difficult ASDs, the incidence of arrhythmias (AV block, atrial fibrillation or flutter), device embolization, embolic events or migraine. A subgroup analysis according to patients age and anatomy of the defect will be performed.

Outlook: The IRFACODE II study is the first trial intended to detect the actual incidence of erosion after ASD closure using the Flex II device. Although the trial is primarily designed to study the safety and device performance, the incidence of other potential side effects will be also evaluated.

ELIGIBILITY:
Inclusion Criteria: ASD for device closure

-

Exclusion Criteria:

* life expectancy < 12 months
* participating in another study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients undergoing interventional ASD closure by using the Occlutech Flex II device
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
number of erosions | minimum 1 year
  detection of erosions of the atrial wall after ASD closure

SECONDARY OUTCOMES:
number of arrhythmias | minimum 1 year
  detection of arrhythmias after ASD closure
successful implantation | minimum 1 year
  number of successful device implantations after device was placed inside the heart
embolization | minimum 1 year
  number of events of device embolization during Implantation and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus A Haas, MD, PhD, Principal Investigator — Ludwig-Maximilians - University of Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haas NA, Soetemann DB, Ates I, Baspinar O, Ditkivskyy I, Duke C, Godart F, Lorber A, Oliveira E, Onorato E, Pac F, Promphan W, Riede FT, Roymanee S, Sabiniewicz R, Shebani SO, Sievert H, Tin D, Happel CM. Closure of Secundum Atrial Septal Defects by Using the Occlutech Occluder Devices in More Than 1300 Patients: The IRFACODE Project: A Retrospective Case Series. Catheter Cardiovasc Interv. 2016 Oct;88(4):571-581. doi: 10.1002/ccd.26497. Epub 2016 Mar 31. PMID 27029396